CLINICAL TRIAL: NCT00376792
Title: An Open Randomized Phase III Trial of Six Cycles of Docetaxel Versus Surveillance After Radical Prostatectomy in High Grade Prostate Cancer Patients With Margin Positive T2 or T3 Tumours
Brief Title: Docetaxel Compared With Observation in Treating Patients Who Have Undergone Radical Prostatectomy for Prostate Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scandinavian Prostate Cancer Group (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000456773; SPCG-12; EUDRACT-2005-002355-40; EU-20638; SANOFI-AVENTIS-SPCG-12; SPCG-ADPRO
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-06

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Watchful Waiting; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: docetaxel
Other: active surveillance
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving docetaxel after surgery may kill any tumor cells that remain after surgery. Sometimes, after surgery, the tumor may not need more treatment until it progresses. In this case, observation may be sufficient. It is not yet known whether giving docetaxel after surgery is more effective than observation in treating prostate cancer.

PURPOSE: This randomized phase III trial is studying docetaxel to see how well it works compared with observation in treating patients who have undergone radical prostatectomy for prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare time to prostate-specific antigen (PSA) progression in patients with margin-positive tumors after undergoing radical prostatectomy for high-grade prostate cancer treated with docetaxel versus observation.

Secondary

* Compare PSA doubling time in patients treated with these regimens.
* Compare quality of life of these patients.
* Compare overall and metastasis-free survival of patients treated with these regimens.

OUTLINE: This is a prospective, open-label, randomized, multicenter study. Patients are stratified according to participating center and tumor stage (pT2 vs pT3). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, directly after and 6 months after completing study treatment, and then annually thereafter.

* Arm II: Patients undergo observation until PSA progression (defined as PSA ≥ 0.5 ng/mL) Quality of life is assessed at baseline, week 19, and annually thereafter.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 396 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate meeting one of the following criteria after undergoing radical prostatectomy:

  * pT2 with Gleason score 4+3 or 8-10 and positive margins in the radical prostatectomy specimen
  * Any pT3a tumor with Gleason score ≥ 4+3
  * pT3b tumor with Gleason score ≥ 7
* Negative lymph nodes at histological examination (N0)
* Patients with a preoperative prostate-specific antigen (PSA) ≥ 10.0 ng/mL should have undergone a lymph node dissection
* Postoperative PSA must be < 0.5 ng/mL
* Considered at high risk for recurrent disease
* No metastatic (M0) disease

  * Negative bone scan

PATIENT CHARACTERISTICS:

* WHO/ECOG performance status 0-1
* Hemoglobin ≥ 11.0 g/dL
* Neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 150,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin normal
* AST and ALT ≤ 1.5 times ULN
* Alkaline phosphatase < 1.5 times ULN
* No active untreated infectious disease (e.g., tuberculosis or methicillin-resistant Staphylococcus aureus)
* No active gastric ulcer
* No known hypersensitivity to polysorbate 80
* No symptomatic peripheral neuropathy ≥ grade 2
* No myocardial infarction within the past 6 months
* No other unstable cardiovascular disease within the past 6 months
* No other serious illness or medical condition
* No altered psychological or physical state that would preclude study compliance
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior hormonal therapy (e.g., luteinizing hormone-releasing hormone analogues and/or antiandrogens) affecting prostate cancer cells
* No prior radiotherapy to the pelvis
* No prior chemotherapy
* More than 6 months since prior systemic corticosteroids
* No other concurrent anticancer therapy or investigational drugs

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2005-10; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Prostate-specific antigen (PSA) progression

SECONDARY OUTCOMES:
PSA doubling time
Quality of Life
Metastasis-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Goran Ahlgren, MD, PhD, Study Chair — Skane University Hospital; Per Flodgren, MD, PhD — Lund University Hospital
Locations (8):
- Denmark (2):
  - Aarhus Universitetshospital - Aarhus Sygehus, Aarhus
  - Copenhagen County Herlev University Hospital, Copenhagen
- Tampere University Hospital, Tampere, Finland
- Landspitalinn University Hospital, Reykjavik, Iceland
- Norway (2):
  - Ullevaal University Hospital, Oslo
  - Norwegian University of Science and Technology, Trondheim
- Sweden (2):
  - Lund University Hospital, Lund
  - Malmo University Hospital, Malmo